CLINICAL TRIAL: NCT06794255
Title: Randomized Controlled Trial on Vitamin C Supolementation for HealthRegulation in Middle-Aged and Elderly Adults
Brief Title: Exploratory Study on the Role of Vitamin C in Promoting Health in Middle-Aged and Elderly Adults
Acronym: VitC-Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: The First Affiliated Hospital of Nanchang University (Other); People's Hospital of Quzhou (Other)
Responsible Party: Principal Investigator, Jie Qiao, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: M2024651; 88888888 (Other Grant/Funding Number: Peking University Third Hospital)
Record Dates: First submitted 2025-01-10; First posted 2025-01-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-01

CONDITIONS: Ageing
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vitamin C (Experimental): Participants will take the synthetic vitamin C twice a day, 500mg per time
  Interventions: Dietary Supplement: Vitamin C
- Placebo (Placebo Comparator): Participants will take tablets with the same texture, flavor, and appearance as the experimental group twice a day, 500mg per time.
  Interventions: Other: Placebo
- Baseline control (No Intervention): Recruit 100 healthy individual volunteers aged 18 - 70 years old (20 volunteers in the age range of 18 - 30, 20 in 30 - 40, 20 in 40 - 50, 20 in 50 - 60, and 20 in 60 - 70, with an equal number of males and females in each age group) as the baseline control for age-related changes. This group will not receive any intervention.

INTERVENTIONS:
Dietary Supplement: Vitamin C — Participants swallow synthetic vitamin C tablets 500mg with water, twice a day.
  Arms: Vitamin C
Other: Placebo — Participants swallow tablets with the same texture, flavor, and appearance as the experimental group 500mg with water, twice a day.
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to understand whether oral vitamin C can help delay the aging of middle-aged and elderly individuals, search for sensitive biomarkers of human aging, and provide new paradigms and scientific guidance for aging intervention with small molecule drugs. The main questions it aims to answer are as follows:

* Can oral vitamin C effectively improve the aging-related indicators?
* What is the safety of participants when taking vitamin C supplements?

Researchers will compare vitamin C with a placebo to observe whether vitamin C is effective in intervening in the aging of middle-aged and elderly individuals. Participants need to:

* Take 2 tablets (250mg/tablet) of vitamin C or placebo after breakfast and dinner every day for 12 consecutive months;
* Go to the designated place for a face-to-face follow-up every 6 months and receive a telephone follow-up every 2 months, and pick up subsequent drugs during the follow-up;
* Honestly inform the medication situation during each follow-up;
* Report any discomfort or adverse reactions that occur during the treatment process to the researchers;
* Fill in a questionnaire about their own health status during each follow-up;
* After 6 months and 12 months of intervention, conduct a comprehensive health examination as required, including blood tests and other items.

ELIGIBILITY:
Inclusion Criteria:

* Age: 55-65 years (for the experimental and control groups) or 18-70 years (for the baseline control group assessing aging changes).
* Health Status: Deemed to be in good health based on medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Weight: BMI within the range of 18.5-28 kg/m².
* Informed Consent: Capable of signing the informed consent form and complying with the requirements and restrictions outlined in the study protocol.

Exclusion Criteria:

* Disease Status:Uncontrolled medical conditions or any disease that, in the investigator's opinion, may pose an inappropriate risk or contraindication or interfere with the study's objectives, conduct, or evaluation.Severe chronic or acute diseases (e.g., cancer, heart failure, renal insufficiency, COPD, diabetes, active liver disease, metabolic acidosis, poorly controlled hypertension, epilepsy, recent cardiovascular events, inflammatory bowel disease, neurological disorders, infectious diseases, severe autoimmune diseases, etc.).
* Weight: BMI < 18.5 or BMI > 28.
* Substance/Alcohol Abuse: Ongoing alcohol or drug abuse, or excessive alcohol consumption.
* Medical History: History of gastrointestinal diseases, hyperuricemia, kidney or urinary tract stones, glucose-6-phosphate dehydrogenase deficiency, or paroxysmal nocturnal hemoglobinuria.
* Allergy: Allergy to vitamin C or any component of its formulation.
* Recent Medication Use: Use of high-dose vitamin C, vitamin E, low-dose aspirin, acarbose, metformin, NMN/NR, or other anti-aging/weight-loss drugs within the past 3 months.
* Informed Consent: Inability to provide informed consent.
* Other: Any physical condition that, in the investigator's opinion, may adversely affect the study process or outcomes.
* Clinical Research Participation: Participation in any other clinical research within 3 months prior to screening or during the study period, or receipt of chemotherapy, radiotherapy, biologic therapy, small-molecule therapeutic agents, or investigational drugs, with incomplete recovery from related side effects (excluding alopecia or potential neuropathy).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of vitamin C in intervening in aging | 12 months
  DNA methylation composite clock

SECONDARY OUTCOMES:
blood cell transcriptomics | 12 months
  blood cell transcriptomics
proteomics | 12 months
  proteomics in blood
metabolomics | 12 months
  metabolomics in blood
gut microbiome | 12 months
  gut microbiome in fecal sample
Cognitive function | 1 year
  Trail Making Test
Physical Fitness Test | 1 year
  The score of Purdue pegboard test, Grip Strength Test，and Single Leg Stand Test with Eyes Closed
Maximal oxygen consumption | 1 year
  Maximal oxygen consumption
Motor Function | 1 year
  Hamilton Anxiety Scale
muscle mass | 1 year
  By means of measurement of lean body mass using dual-energy X-ray absorptiometry (DXA)
Cardiovascular disease | 1 year
  Standardised composite score (Z score) of systolic blood pressure, LDL cholesterol, and body-mass index (BMI).
Vitamin C level | 1 year
  Vitamin C level in serum

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The first affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - People's Hospital of Quzhou, Quzhou, Zhejiang
  - Peking University Third Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No
I have decided not to share the IPD from this study due to concerns about participant privacy and confidentiality. Our study will include multiple-omic data, including genomic data. There are legal and ethical considerations that restrict the sharing of sensitive health information and genetic information without consent. Furthermore, the resources required to prepare and manage the data for external sharing are currently beyond our capacity. Therefore, to ensure the protection of our participants and comply with ethical standards, we have opted not to share the IPD at this time.